CLINICAL TRIAL: NCT05023863
Title: The Effect of Alpha Lipoic Acid on the Incidence and Severity of Radiotherapy-Induced Oral Mucositis in Head and Neck Cancer Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Bishoy Anwar, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PHLCLINICAL
Record Dates: First submitted 2021-08-01; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Radiation-Induced Mucositis
Keywords: Head and Neck cancer; Alpha Lipoic Acid; Mucositis
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis | interventions — Thioctic Acid; Radiation

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, controlled, single blinded study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alpha Lipoic Acid Group (intervention group) (Active Comparator): 35 patients will receive radiation therapy with or without platinum-based chemotherapy in addition to alpha lipoic acid 600 mg tablets twice daily (throughout the radiotherapy period). .
  Interventions: Drug: Alpha Lipoic Acid 600 MG Oral Tablets; Radiation: radiation or concurrent chemoradiation
- Control Group (Placebo Comparator): 35 Patients will receive radiation therapy with or without platinum-based chemotherapy in addition to placebo tablets twice daily (throughout the radiotherapy period)
  Interventions: Other: Placebo tablets; Radiation: radiation or concurrent chemoradiation

INTERVENTIONS:
Drug: Alpha Lipoic Acid 600 MG Oral Tablets — Alpha Lipoic Acid (ALA) is a drug which has been used in treatment of diabetic neuropathy . It act through enhancing nitric oxide-mediated endothelium-dependent vasodilation, thus improving microcirculation in patients with diabetic polyneuropathy. It is considered a safe drug, generally with a daily dose of 200 to 2400 mg/day is considered tolerable without significant side effects. Only gastrointestinal tracts side effects like nausea, vomiting, dyspepsia and abdominal pain have been described in some clinical trials. Also FDA experts confirm its safety and efficacy in humans
  Arms: Alpha Lipoic Acid Group (intervention group)
Other: Placebo tablets — placebo tablets of the same generic of active drug which contain all the same ingredients as active tablets except alpha lipoic acid
  Arms: Control Group
Radiation: radiation or concurrent chemoradiation — radiation or concurrent radiotherapy plus platinum-based chemotherapy

SUMMARY:
A prospective, randomized, controlled, single-blinded study will be conducted at Clinical Oncology department, Ain Shams University Hospitals, assessing the effect of Alpha Lipoic Acid on the incidence and severity of radiotherapy induced oral mucositis in Head and Neck cancer patients.

DETAILED DESCRIPTION:
All patients presenting to the Clinical Oncology department, Ain Shams University Hospitals, will be assessed for eligibility as follow:

Inclusion criteria:

* Age >18 years.
* Diagnosis of stage I, II, III or IV squamous cell carcinoma, nasopharyngeal carcinoma.
* Measurable disease on CT scan at baseline.
* Planned to receive radiotherapy with a total dose 60 grays or more divided on 30 fractions with or without cisplatin (100 mg/m2, administered intravenously every 21 days for three cycles or 40 mg/m2 administered weekly for up to 7 weeks).
* Adequate liver function (liver transaminases level < 3 times upper normal limits and total bilirubin < 1.5 times upper normal limits).
* Adequate kidney function (estimated glomerular filtration rate >60 ml/min).
* Adequate bone marrow function (WBCs count > 3000 cells/mm3, ANC count >1500 cells/mm3 and platelets count > 100,000 cells/mm3).

Exclusion criteria:

Patients will be excluded if they have any of the following:

* Diagnosis of Thyroid cancer.
* Presence of other primary cancers.
* Treatment with alpha lipoic acid for any other indication.
* Allergy to alpha lipoic acid.
* Pregnant or lactating women. Eligible patients will be randomized to either… Alpha Lipoic Acid Group (intervention group): 35 patients will receive radiation therapy with or without platinum-based chemotherapy in addition to alpha lipoic acid 600 mg tablets twice daily (throughout the radiotherapy period). The medication will be brought from EVA company ( an Egyptian drug company ) under the trade name of thiotacid 600 mg tablets.

Control Group: 35 Patients will receive radiation therapy with or without platinum-based chemotherapy plus placebo tablets of thiotacid throughout the radiation period

All patients will be followed up weekly to assess the incidence and severity of radiation induced oral mucositis using the radiotherapy oncology group criteria also blood samples will be drawn at baseline , after three weeks (middle of radiation period) at the end of radiation period to asses changes in CRP and TAC levels

ELIGIBILITY:
Inclusion Criteria:

* • Age >18 years.

  * Diagnosis of stage I, II, III or IV squamous cell carcinoma, nasopharyngeal carcinoma.
  * Measurable disease on CT scan at baseline.
  * Planned to receive radiotherapy with a total dose 60 grays or more divided on 30 fractions with or without cisplatin (100 mg/m2, administered intravenously every 21 days for three cycles or 40 mg/m2 administered weekly for up to 7 weeks).
  * Adequate liver function (liver transaminases level < 3 times upper normal limits and total bilirubin < 1.5 times upper normal limits).
  * Adequate kidney function (estimated glomerular filtration rate >60 ml/min).
  * Adequate bone marrow function (WBCs count > 3000 cells/mm3, ANC count >1500 cells/mm3 and platelets count > 100,000 cells/mm3).

Exclusion Criteria:

* ● Diagnosis of Thyroid cancer.

  * Presence of other primary cancers.
  * Treatment with alpha lipoic acid for any other indication.
  * Allergy to alpha lipoic acid.
  * Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of radiation induced oral mucositis | 4 months
  The patients will be followed up during the whole period of radiation and up to six weeks after radiation to evaluate the incidence and severity of radiation induced mucositis. Severity will be assessed by the oncologist using radiotherapy oncology group criteria (RTOG criteria)

SECONDARY OUTCOMES:
Time to develop grade III or IV radiation induced oral mucositis: | 4 months
  For each patient, the time from the start of radiotherapy till the development of grade III or IV RIOM will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Abdan M. Alfa-lipoic acid controls tumor growth and modulates hepatic redox state in Ehrlich-ascites-carcinoma-bearing mice. ScientificWorldJournal. 2012;2012:509838. doi: 10.1100/2012/509838. Epub 2012 May 1. PMID 23002387
- [Background] Bloomer WD, Hellman S. Normal tissue responses to radiation therapy. N Engl J Med. 1975 Jul 10;293(2):80-3. doi: 10.1056/NEJM197507102930206. No abstract available. PMID 1093032
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Elsabagh HH, Moussa E, Mahmoud SA, Elsaka RO, Abdelrahman H. Efficacy of Melatonin in prevention of radiation-induced oral mucositis: A randomized clinical trial. Oral Dis. 2020 Apr;26(3):566-572. doi: 10.1111/odi.13265. Epub 2020 Jan 15. PMID 31869853
- [Background] Gillison ML. Human papillomavirus-related diseases: oropharynx cancers and potential implications for adolescent HPV vaccination. J Adolesc Health. 2008 Oct;43(4 Suppl):S52-60. doi: 10.1016/j.jadohealth.2008.07.002. PMID 18809146
- [Background] Jung JH, Jung J, Kim SK, Woo SH, Kang KM, Jeong BK, Jung MH, Kim JH, Hahm JR. Alpha lipoic acid attenuates radiation-induced thyroid injury in rats. PLoS One. 2014 Nov 17;9(11):e112253. doi: 10.1371/journal.pone.0112253. eCollection 2014. PMID 25401725
- [Background] Kim H, Yoo WS, Jung JH, Jeong BK, Woo SH, Kim JH, Kim SJ. Alpha-Lipoic Acid Ameliorates Radiation-Induced Lacrimal Gland Injury through NFAT5-Dependent Signaling. Int J Mol Sci. 2019 Nov 13;20(22):5691. doi: 10.3390/ijms20225691. PMID 31766286
- [Background] Kim JH, Jeong BK, Jang SJ, Yun JW, Jung MH, Kang KM, Kim TG, Woo SH. Alpha-Lipoic Acid Ameliorates Radiation-Induced Salivary Gland Injury by Preserving Parasympathetic Innervation in Rats. Int J Mol Sci. 2020 Mar 25;21(7):2260. doi: 10.3390/ijms21072260. PMID 32218158
- [Background] Kusiak A, Jereczek-Fossa BA, Cichonska D, Alterio D. Oncological-Therapy Related Oral Mucositis as an Interdisciplinary Problem-Literature Review. Int J Environ Res Public Health. 2020 Apr 3;17(7):2464. doi: 10.3390/ijerph17072464. PMID 32260309
- [Background] Logan RM, Stringer AM, Bowen JM, Gibson RJ, Sonis ST, Keefe DM. Serum levels of NFkappaB and pro-inflammatory cytokines following administration of mucotoxic drugs. Cancer Biol Ther. 2008 Jul;7(7):1139-45. doi: 10.4161/cbt.7.7.6207. Epub 2008 Apr 29. PMID 18535404
- [Background] Lott IT, Doran E, Nguyen VQ, Tournay A, Head E, Gillen DL. Down syndrome and dementia: a randomized, controlled trial of antioxidant supplementation. Am J Med Genet A. 2011 Aug;155A(8):1939-48. doi: 10.1002/ajmg.a.34114. Epub 2011 Jul 7. PMID 21739598
- [Background] Mallick S, Benson R, Rath GK. Radiation induced oral mucositis: a review of current literature on prevention and management. Eur Arch Otorhinolaryngol. 2016 Sep;273(9):2285-93. doi: 10.1007/s00405-015-3694-6. Epub 2015 Jun 27. PMID 26116012
- [Background] Marur S, Forastiere AA. Head and Neck Squamous Cell Carcinoma: Update on Epidemiology, Diagnosis, and Treatment. Mayo Clin Proc. 2016 Mar;91(3):386-96. doi: 10.1016/j.mayocp.2015.12.017. PMID 26944243
- [Background] Moreira PI, Harris PL, Zhu X, Santos MS, Oliveira CR, Smith MA, Perry G. Lipoic acid and N-acetyl cysteine decrease mitochondrial-related oxidative stress in Alzheimer disease patient fibroblasts. J Alzheimers Dis. 2007 Sep;12(2):195-206. doi: 10.3233/jad-2007-12210. PMID 17917164
- [Background] Pearman TP, Beaumont JL, Paul D, Abernethy AP, Jacobsen PB, Syrjala KL, Von Roenn J, Cella D. Evaluation of treatment- and disease-related symptoms in advanced head and neck cancer: validation of the national comprehensive cancer network-functional assessment of cancer therapy-head and neck cancer symptom index-22 (NFHNSI-22). J Pain Symptom Manage. 2013 Jul;46(1):113-20. doi: 10.1016/j.jpainsymman.2012.06.004. Epub 2012 Sep 25. PMID 23017622
- [Background] Reljanovic M, Reichel G, Rett K, Lobisch M, Schuette K, Moller W, Tritschler HJ, Mehnert H. Treatment of diabetic polyneuropathy with the antioxidant thioctic acid (alpha-lipoic acid): a two year multicenter randomized double-blind placebo-controlled trial (ALADIN II). Alpha Lipoic Acid in Diabetic Neuropathy. Free Radic Res. 1999 Sep;31(3):171-9. doi: 10.1080/10715769900300721. PMID 10499773
- [Background] Sayed R, El Wakeel L, Saad AS, Kelany M, El-Hamamsy M. Pentoxifylline and vitamin E reduce the severity of radiotherapy-induced oral mucositis and dysphagia in head and neck cancer patients: a randomized, controlled study. Med Oncol. 2019 Nov 21;37(1):8. doi: 10.1007/s12032-019-1334-5. PMID 31748905
- [Background] Siddiqui F, Movsas B. Management of Radiation Toxicity in Head and Neck Cancers. Semin Radiat Oncol. 2017 Oct;27(4):340-349. doi: 10.1016/j.semradonc.2017.04.008. PMID 28865517
- [Background] Sonis ST. Pathobiology of oral mucositis: novel insights and opportunities. J Support Oncol. 2007 Oct;5(9 Suppl 4):3-11. PMID 18046993
- [Background] Ziegler D, Nowak H, Kempler P, Vargha P, Low PA. Treatment of symptomatic diabetic polyneuropathy with the antioxidant alpha-lipoic acid: a meta-analysis. Diabet Med. 2004 Feb;21(2):114-21. doi: 10.1111/j.1464-5491.2004.01109.x. PMID 14984445